CLINICAL TRIAL: NCT05610605
Title: Randomized Clinical Trial to Assess the Efficacy of an Educational Programme for Prevention and Treatment of Frailty in Older Adults Living in the Community: FRAGSALUD Programme
Brief Title: Education for Prevention and Treatment of Frailty
Acronym: FRAGSALUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Collaborators: University of Malaga (Other); Instituto de investigación e innovación biomédica de Cádiz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FRAGSALUD
Record Dates: First submitted 2022-02-09; First posted 2022-11-09 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2022-02

CONDITIONS: Frailty; Frail Elderly Syndrome
Keywords: Elderly Persons; Aging; Cost-Efficiency Analysis; Health Education
MeSH Terms: conditions — Frailty; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants who do not receive attention from the Fragsalud program. The control group follows the usual care and preventive measures in Primary Care, according to different protocols implemented and the criteria of nurses and family doctors responsible for their care.
- Intervention Group (Experimental): The FRAGSALUD Programme is a multidomain intervention programme, which covers the prevention and treatment of frailty from different aspects, fundamentally from a physical and cognitive aspect and to maintain social integration, although other modifiable factors that are related to the presence of fragility such as hearing impairment, visual deficit or depression.
  Interventions: Other: Health intervention programme: FRAGSALUD

INTERVENTIONS:
Other: Health intervention programme: FRAGSALUD — The FRAGSALUD Program consists in two parts, a first part of health education that will be taught in a group in four sessions, and a second part of individual treatment and follow-up, individual consultations will have a bimonthly periodicity until reaching one year, at which time that the program ends and a final evaluation will be carried out to assess whether the changes are maintained 15 months after the start.
  Arms: Intervention Group

SUMMARY:
Frailty is a condition with a high prevalence in older adults, leading to higher vulnerability and increasing the risk of adverse health outcomes and disabilities. The aging of the population in Spain is accelerating quickly, consequently, it is necessary to advise the population on the appropriate path to healthy aging, free of fragility and their secondary problems.

DETAILED DESCRIPTION:
To evaluate the efficacy and efficiency of a Fragsalud program for the prevention and multifactorial treatment of frailty in people over 65 years of age living in the community compared to the usual treatment. Material and methods: A Single blind randomized, two-arm clinical trial; control group and intervention group, multicenter, with 15 months of follow-up, with evaluations blinded at the beginning, and in the follow-up at 12 and 15 months. A recruitment of 196 people over 65 years of age with criteria of pre-frailty or frailty according to Fried's criteria. The Fragsalud education program will be taught in the intervention group; while control group will follow the usual health care. The evolution of the criteria of frailty, cognitive state, eating pattern, emotional state, quality of sleep, perceived social support, quality of life, functional capacity in daily life, adverse results, assessment of self-efficacy and cost-utility analysis variables will be evaluated. Possible confounding factors such as sociodemographic variables, comorbidity and polymedication will be controlled. Intention-to-treat analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years of age who present frailty or pre-frailty, assessed using the Fried criteria adapted to Spanish population;
* Patients belonging to Clinical Management Units participating in the study and who will remain in it for the 15 months of the study;
* Patients who can come to the Health Center alone or accompanied.

Exclusion Criteria:

* Patients with no full control of their capabilities.
* Patients who do not understand Spanish;
* Patients with allergies to plastic or metal.
* Patients who are instutionalized.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 235 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: María Ángeles Vázquez Sanchez, PhD, Principal Investigator — Universidad de Málaga
Locations (1):
- Faculty of Education, Puerto Real, Cádiz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez-Mariscal A, Corral-Perez J, Vazquez-Sanchez MA, Avila-Cabeza-de-Vaca L, Costilla M, Casals C. Benefits of an educational intervention on functional capacity in community-dwelling older adults with frailty phenotype: A randomized controlled trial. Int J Nurs Stud. 2025 Feb;162:104955. doi: 10.1016/j.ijnurstu.2024.104955. Epub 2024 Nov 9. PMID 39579605
- [Derived] Corral-Perez J, Vazquez-Sanchez MA, Casals-Sanchez JL, Contreras-Garcia FJ, Costilla M, Casals C. A 6-month educational program improves sleep behaviour in community-dwelling frail older adults: A randomised controlled trial. Sleep Med. 2024 Sep;121:196-202. doi: 10.1016/j.sleep.2024.07.011. Epub 2024 Jul 10. PMID 39002328
- [Derived] Casals C, Corral-Perez J, Avila-Cabeza-de-Vaca L, Gonzalez-Mariscal A, Carrion-Velasco Y, Rodriguez-Martinez MC, Jimenez-Cebrian AM, Vazquez-Sanchez MA. Exploring the interplay of frailty, physical function, physical activity, nutritional status, and their association with quality of life and depressive symptoms in older adults with the frailty phenotype. Int J Geriatr Psychiatry. 2024 Mar;39(3):e6078. doi: 10.1002/gps.6078. PMID 38470426
- [Derived] Corral-Perez J, Casals C, Avila-Cabeza-de-Vaca L, Gonzalez-Mariscal A, Mier A, Espinar-Toledo M, Garcia-Agua Soler N, Vazquez-Sanchez MA. Associations Between Physical Activity and Inactivity Levels on Physical Function and Sleep Parameters of Older Adults With Frailty Phenotype. J Appl Gerontol. 2024 Jul;43(7):910-921. doi: 10.1177/07334648231218095. Epub 2023 Dec 1. PMID 38038169

RESULTS

PARTICIPANT FLOW:
Period: 6-month Assessment
Arm/Group | Control Group | Intervention Group
Started | 117 | 118
Completed | 95 | 115
Not Completed | 22 | 3
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 20 | 0
Not completed — Institutionalized | 1 | 2
Period: 12-month Assessment
Arm/Group | Control Group | Intervention Group
Started | 95 | 115
Completed | 90 | 109
Not Completed | 5 | 6
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 1 | 4
Not completed — Institutionalized | 2 | 1

BASELINE CHARACTERISTICS:
Population: The study enrolled individuals residing in the community across Cadiz and Malaga pronvices. To meet the criteria for participation, individuals needed to be aged 65 years or above, display at least one aspect of Fried's frailty phenotype and being in full possession of their faculties to voluntarily participate in the study. Those ineligible for participation encompassed individuals in institutional settings, and individuals categorized as robust (without any Fried's frailty criteria).
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Total
Number analyzed (Participants) | 117 | 118 | 235
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.6 (6.4) | 73.2 (6.0) | 74.4 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 95 | 159
  Male | 53 | 23 | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 117 | 118 | 235
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 117 | 118 | 235
Fried's Frailty Criteria [Mean (Standard Deviation); unit: scores on a scale] — Assessment of frailty using the Fried Frailty Phenotype. This is a five-component measure used to classify frailty status (unintentional weight loss, exhaustion, weakness, slow walking speed, and low physical activity).
  A score of 1 is assigned for each criterion met, yielding a total score that ranges from 0 to 5. A higher score indicates a worse outcome (greater frailty).
  0 = Robust (non-frail)
  1-2 = Pre-frail
  3-5 = Frail
  scores on a scale | 2.0 (0.9) | 2.1 (1.0) | 2.1 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the Change of Baseline Fried Frailty Criteria at 6 Months
Description: Assessment of frailty using the Fried Frailty Phenotype. This is a five-component measure used to classify frailty status (unintentional weight loss, exhaustion, weakness, slow walking speed, and low physical activity).
  A score of 1 is assigned for each criterion met, yielding a total score that ranges from 0 to 5. A higher score indicates a worse outcome (greater frailty).
  0 = Robust (non-frail)
  1-2 = Pre-frail
  3-5 = Frail
Time Frame: Preintervention/Postintervention (0 and 6 months)
Population: Older adults (>65 years) with frailty phenotype
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 95 | 115
scores on a scale | 2.3 (1.1) | 1.4 (0.9)

2. Primary Outcome: Evaluation of the Change of Baseline Fried Frailty Criteria at 12 Months
Description: as for outcome 1
Time Frame: Preintervention/Retest (0 and 12 months)
Population: Older adults (>65 years) with frailty phenotype.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 90 | 109
scores on a scale | 2.5 (1.2) | 1.4 (1.0)

ADVERSE EVENTS:
Time Frame: The data was obtained at the end of the intervention (6 months) and 6 months after the completion of the intervention (12 months)
Description: Adverse events were systematically assessed by study personnel at the 6-month and 12-month follow-up visits. All-cause mortality was tracked for all participants.
Arm/Group | Control Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 3/117 | 2/118
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/118
Other Adverse Events (participants affected / at risk) | 0/117 | 0/118

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-24): https://cdn.clinicaltrials.gov/large-docs/05/NCT05610605/Prot_SAP_000.pdf